CLINICAL TRIAL: NCT06171152
Title: Examining the Utility of GLP-1 Agonists as Neuroprotective Agents Through a Pilot Clinical Trial in High Risk Population With Neurocognitive Deficits and Obesity
Brief Title: Study of Liraglutide (A Weight Loss Drug) in High Risk Obese Participants With Cognitive and Memory Issues
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-0848
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis; Long COVID; Long Covid19; Obese; Obesity; Obesity, Morbid; Acute Leukemia in Remission
MeSH Terms: conditions — Multiple Sclerosis; Post-Acute COVID-19 Syndrome; Obesity; Obesity, Morbid | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group 1 (Drug Regimen A) (Experimental): During the study, liraglutide will be given in "cycles." A cycle is a scheduled period of time for taking study drugs. For this study, each cycle length as well as the dose of liraglutide participants take will be based on the drug regimen (or schedule) they receive. The drug regimen receive each participant receives will be selected using a random assignment process, similar to flipping a coin.
  Participants in this study group will receive Drug Regimen A, which means they will take liraglutide at the below doses and times:
  Dose Schedule Cycle Length 0.6mg Daily 1 week 1.2mg Daily 1 week 1.8mg Daily 1 week 2.4mg Daily 1 week 3.0mg Daily 8 weeks
  Interventions: Drug: Liraglutide Pen Injector [Saxenda]; Other: Medication Diary
- Study Group 2 (Drug Regimen B) (Experimental): During the study, liraglutide will be given in "cycles." A cycle is a scheduled period of time for taking study drugs. For this study, each cycle length as well as the dose of liraglutide participants take will be based on the drug regimen (or schedule) they receive. The drug regimen receive each participant receives will be selected using a random assignment process, similar to flipping a coin.
  Participants in this study group will receive Drug Regimen B, which means they will take liraglutide at the below doses and times:
  Dose Schedule Cycle Length 0.6mg Daily 5 weeks 1.2mg Daily 1 week 1.8mg Daily 1 week 2.4mg Daily 1 week 3.0mg Daily 4 weeks
  Interventions: Drug: Liraglutide Pen Injector [Saxenda]; Other: Medication Diary

INTERVENTIONS:
Drug: Liraglutide Pen Injector [Saxenda] — A weight loss drug that can be taken at home. Liraglutide will be provided as an injectable pen that participants can inject in the stomach, thigh or upper arm. A member of the research team will give you instructions on how to inject liraglutide using the injectable pen and answer any questions.
  Other Names: Saxenda; Victoza
Other: Medication Diary — Participants will be asked to maintain a medication diary of each dose of liraglutide. A member of the research team will provide a copy of this diary for participants to complete. Participants will be asked to return this medication diary to research staff at each clinic visit.

SUMMARY:
This study is for people who have multiple sclerosis, acute leukemia (in remission), or long-COVID and a Body Mass Index over 27 and may struggle with cognitive issues such as remembering information, concentrating, or making decisions that affect everyday life.

By doing this study, researchers hope to learn how liraglutide (Saxenda®), a weight loss drug, affects levels of a certain disease marker in the body called Brain Derived Neurotrophic Factor (BDNF). Participation in this research will last about 21 weeks.

DETAILED DESCRIPTION:
This study is for people who have multiple sclerosis, acute leukemia (in remission), or long-COVID and a Body Mass Index over 27 and may struggle with cognitive issues such as remembering information, concentrating, or making decisions that affect everyday life. By doing this study, researchers hope to learn how liraglutide (Saxenda®), a weight loss drug, affects levels of a certain disease marker in the body called Brain Derived Neurotrophic Factor (BDNF).

Previous research has shown that liraglutide may help regulate BDNF levels, which can be linked to issues with cognitive and mental performance. Participation in this research will last about 21 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MS, acute leukemia in remission, or long-COVID and subjective symptoms of cognitive impairment a. Patients with acute leukemia must be in remission for at least 6 months but may be on maintenance therapy

   * Must have BMI greater than or equal to 27 along with one weight related condition such as hypertension, insulin resistance, or dyslipidemia or with BMI greater than or equal to 30 alone
   * Ages ≥18 but <40 years old
   * Adequate organ function as defined by the following:

     1. Creatinine ≤1.5 mg/dL
     2. Aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤5 x upper limit normal (ULN) and bilirubin ≤1.5 mg/dL
   * Participants must be at least 2 months from major surgery, radiation therapy, or participation in other investigational trials, and must have recovered from clinically significant toxicities related to these prior treatments.
   * Female participants of childbearing potential must have negative results for a pregnancy test at baseline testing time point
   * Must be willing to use appropriate contraception
   * The effects of liraglutide on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 8 weeks after completion of liraglutide administration.
   * Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of multiple endocrine neoplasia type 2 (MEN2)
* Personal or family history of thyroid cancer
* Previous or current diagnosis of acute and/or chronic pancreatitis
* Any prior GLP-1 agonist therapy
* Poorly controlled diabetes mellitus with an indication for liraglutide (Victoza) for its management
* Previous or current diagnosis of fibromyalgia
* Participants who are receiving any other investigational agents.
* Participants with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥ 3 years.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to liraglutide.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because liraglutide is a Category X agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with liraglutide, breastfeeding should be discontinued prior to enrollment in the trial.
* Participants with congenital cognitive dysfunction or severe cognitive dysfunction unrelated to diagnosis of leukemia, Multiple Sclerosis, or COVID.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Serum Brain Derived Neurotrophic Factor (BDNF) after 8 Weeks | 8 weeks
  Change from baseline in serum Brain Derived Neurotrophic Factor (BDNF) levels after reaching the goal dose of GLP-1 agonist (8 weeks).

SECONDARY OUTCOMES:
Change from Baseline in Serum Brain Derived Neurotrophic Factor (BDNF) after 4 Weeks | 4 weeks
  Change from baseline in serum Brain Derived Neurotrophic Factor (BDNF) levels at 4 weeks.
Change from Baseline in Serum Brain Derived Neurotrophic Factor (BDNF) after 12 Weeks | 12 weeks
  Change from baseline in serum Brain Derived Neurotrophic Factor (BDNF) levels at 12 weeks.
Change from Baseline in Serum Brain Derived Neurotrophic Factor (BDNF) after 21 Weeks | 21 weeks
  Change from baseline in serum Brain Derived Neurotrophic Factor (BDNF) levels at discontinuation of study drug (21 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Adam DuVall, MD, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF